CLINICAL TRIAL: NCT02328911
Title: Laser Therapy Treatment of Peripheral Neuropathic Pain in Individuals With Diabetes
Brief Title: Laser Therapy for Diabetic Peripheral Neuropathic Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruiting qualified subjects.
Sponsor: University of Miami (Other)
Collaborators: LiteCure LLC (Industry)
Responsible Party: Principal Investigator, John E. Lewis, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110921
Record Dates: First submitted 2014-11-16; First posted 2014-12-31 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser treatment (Experimental): Twice-per-week laser treatment for 4 weeks and once-per-week laser treatment for 8 weeks. Inflammatory markers, functional status, and quality of life will be examined.
  Interventions: Device: Laser treatment
- Sham treatment (Sham Comparator): Twice-per-week sham treatment for 4 weeks and once-per-week sham treatment for 8 weeks. Inflammatory markers, functional status, and quality of life will be examined.
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: Laser treatment — Laser energy will be applied to the skin of the back and feet manually by physician though a device with a movable head, in contact with the skin, that emits therapeutic dual-wavelength infrared laser energy as well as red visible light.
  Other Names: LiteCure™ LCT-1000 laser
  Arms: Laser treatment
Device: Sham treatment — A sham treatment will be applied to the skin of the back and feet manually by physician though a device with a movable head, in contact with the skin, that emits only red visible light.
  Other Names: LiteCure™ LCT-1000 laser with laser device disabled
  Arms: Sham treatment

SUMMARY:
The proposed study is a randomized, double-blinded clinical trial to evaluate the efficacy of a course of laser therapy on peripheral neuropathic pain in persons with diabetes. The hypothesis is that laser therapy will produce significant improvement on measures of self-reported pain among adults with diabetes.

DETAILED DESCRIPTION:
The proposed study is a randomized, double-blinded clinical trial to evaluate the efficacy of a course of laser therapy on peripheral neuropathic pain in persons with diabetes. Participants will be assessed at baseline, post-intervention, and 3-months followup, and the study will consist of two treatment arms, including: (a) twice-per-week laser treatment for 4 weeks and once-per-week laser treatment for 8 weeks or (b) same treatment schedule sham (or placebo) for 12 weeks. Additionally, the study will examine inflammatory markers, functional status, and quality of life.

Specific Aim 1. Change from baseline in self-reported pain in a sample of adults with diabetes at their last visit and at 3 months. Hypothesis 1: The laser therapy will produce significant improvement at post-intervention and three-month followup on measures of self-reported pain among adults with diabetes. Specific Aim 2: Decrease biochemical markers of inflammation by investigating levels of cytokines. Hypothesis 2: The laser therapy will produce significant improvement at post-intervention and three-month followup on levels of inflammatory markers.Specific Aim 3: Improve quality of life. Hypothesis 3: The laser therapy will produce significant improvement at post-intervention and three-month followup on quality of life.No substantial psychological, medical, or social risks exist to the participants, other than minor discomfort associated with the venipuncture.

Although all measures to protect confidentiality will be put in place, the possibility exists that electronic data could be jeopardized. In the remote case that such event occurs, it will be immediately reported to the IRB.The proper use of the LiteCure LightForce FX Therapy Laser class IV laser therapy device should be harmless and presents no different risks than similar laser therapy devices currently on the market. At the time of this submission, no serious adverse events have been reported to the company or the regulatory authority by consumers. All study personnel will complete detailed training in the use of the device and will follow the directions of the manufacturer for operating the device; all instructions for use of the device will be followed for each subject.

As reported by LiteCure Medical the LiteCure LightForce FX therapy laser device has been cleared by the FDA, tested according IEC electrical safety standards for medical devices, and manufactured in an ISO13485 compliant facility. These certifications ensure that LiteCure Medical devices are manufactured in state of the art facilities, under strict quality control, and environmental protection standards. Participants will incur no additional appreciable psychological or social risks by participating in this study. The process of interviewing during the assessment may cause discomfort. Discomfort or fatigue may also be experienced in completing the assessment battery.

The information obtained in this study will help in determining the efficacy of using a class IV laser therapy device for neuropathic pain, inflammation, and quality of life in persons with diabetic distal symmetric peripheral neuropathy. By participating in the study, subjects may feel less pain, have lower inflammation, and experience improved quality of life. The minimal risk of participating in this study is reasonable because of the potential benefit gained in pain status, inflammatory status, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Is age 18 or older
2. Has diabetes
3. Has chronic, unresolved neuropathic pain of the feet for more than 3 months
4. able to attend the treatment schedule on-campus for the period of the intervention
5. Is willing to provide informed consent to participate in study

Exclusion Criteria:

1. Has any chronic open wounds on your back or bottom of the feet
2. Is pregnant
3. Diagnosed with schizophrenia, other psychotic disorders, bipolar disorder, major depression with psychotic features, delirium, or alcohol or substance abuse/dependence
4. Diagnosed with a bleeding disorder
5. Diagnosed with aphasia or sensory, motor, or visual disturbances that could interfere with assessments
6. Diagnosed with any major pulmonary, renal, thyroid, hepatic, gastrointestinal, or seizure conditions
7. Had any hematologic or ontological disorders treated with chemotherapy in the previous two years
8. Is currently undergoing any chemotherapy or radiation treatment for cancer
9. Has had more than three major medical or psychiatric hospitalizations in the past year
10. Has been diagnosed with a terminal illness
11. Is you currently participating in another trial with drugs, dietary supplements, or medical treatment that affects neuropathic pain
12. Is currently taking any opioid or other pain medication
13. Is currently taking any pain-relieving nutritional supplement, herb, antioxidants or integrative medicine for diabetic neuropathy
14. Is currently taking prescription or over-the-counter pain relievers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in self-reported pain. | Baseline, from baseline up to 12 weeks (weekly) , and 3-month follow-up.
  Pain will be quantitatively assessed through the use of the vibration testing technique (on-off method) and the Semmes-Weinstein monofilament test .The assessment will be carried out at baseline, baseline up to 12 weeks (weekly), and at 3 months follow-up. In addition, changes in pain over the course of the study will be assessed with several questionnaires and tests, including the Visual Analogue Scale Quadruple Pain Scale, (VAS-QPS), the Neuropathic Pain Scale (NPS), and the Pain Disability Questionnaire (PDQ).

SECONDARY OUTCOMES:
Change in inflammation by measuring levels of biochemical markers. | Baseline, from baseline up to 12 weeks (weekly) , and 3-month follow-up.
  Subjects will have blood drawn, and the tests will include a cytokine panel to check for inflammation in the body at baseline, baseline up to 12 weeks (weekly), and at 3 months follow-up.
Change in quality of life. | Baseline, from baseline up to 12 weeks (weekly) , and 3-month follow-up.
  Subjects will be asked to complete the Medical Outcomes Study Short Form 36 (SF-36) in order to assess the subjects' functional status and measure general health-related quality of life at baseline, baseline up to 12 weeks (weekly), and at 3 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: John E. Lewis, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Clinical Research Building, Department of Psychiatry & Behavioral Sciences, Miami, Florida, United States

REFERENCES:
- [Background] Alster TS, Bryan H, Williams CM. Long-pulsed Nd:YAG laser-assisted hair removal in pigmented skin: a clinical and histological evaluation. Arch Dermatol. 2001 Jul;137(7):885-9. PMID 11453807
- [Background] Hegedus B, Viharos L, Gervain M, Galfi M. The effect of low-level laser in knee osteoarthritis: a double-blind, randomized, placebo-controlled trial. Photomed Laser Surg. 2009 Aug;27(4):577-84. doi: 10.1089/pho.2008.2297. PMID 19530911
- [Background] Kaviani A, Djavid GE, Ataie-Fashtami L, Fateh M, Ghodsi M, Salami M, Zand N, Kashef N, Larijani B. A randomized clinical trial on the effect of low-level laser therapy on chronic diabetic foot wound healing: a preliminary report. Photomed Laser Surg. 2011 Feb;29(2):109-14. doi: 10.1089/pho.2009.2680. Epub 2011 Jan 9. PMID 21214368
- [Background] Meireles SM, Jones A, Jennings F, Suda AL, Parizotto NA, Natour J. Assessment of the effectiveness of low-level laser therapy on the hands of patients with rheumatoid arthritis: a randomized double-blind controlled trial. Clin Rheumatol. 2010 May;29(5):501-9. doi: 10.1007/s10067-009-1347-0. Epub 2010 Jan 16. PMID 20082104
- [Background] Montes-Molina R, Madronero-Agreda MA, Romojaro-Rodriguez AB, Gallego-Mendez V, Prados-Cabiedas C, Marques-Lucas C, Perez-Ferreiro M, Martinez-Ruiz F. Efficacy of interferential low-level laser therapy using two independent sources in the treatment of knee pain. Photomed Laser Surg. 2009 Jun;27(3):467-71. doi: 10.1089/pho.2008.2315. PMID 19405858
- [Background] Moritz AR. Studies of Thermal Injury: III. The Pathology and Pathogenesis of Cutaneous Burns. An Experimental Study. Am J Pathol. 1947 Nov;23(6):915-41. No abstract available. PMID 19970971
- [Background] Naeser MA. Photobiomodulation of pain in carpal tunnel syndrome: review of seven laser therapy studies. Photomed Laser Surg. 2006 Apr;24(2):101-10. doi: 10.1089/pho.2006.24.101. PMID 16706688